CLINICAL TRIAL: NCT05846217
Title: Bell's Palsy With a Duration of Greater Than 8 Weeks Treated With Multiwave Locked System Intervention: A Randomized Controlled Trial
Brief Title: Bell's Palsy With a Duration of Greater Than 8 Weeks Treated With Multiwave Locked System Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Laser-Bell-2023
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Laser Treatment Relieve Symptoms of Chronic Bell's Palsy
Keywords: Bell'palsy; photobiomodulation; RCT; ENoG; EMG

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PBMT Group (Experimental): In PBMT group, we choose 9 points on the affected face, include Mastoid, Preauricular, Temple, Frontalis muscle, Zygomatic muscle, Buccinator muscle, Masseter, Orbicularis oris and Depressor angulli oris. Based on clinical experience, we choose 7 acupoints, including LI4 (HeGu), LI11(QuChi), ST25 (TianShu), ST36 (ZuSanLi), SP6 (SanYinJiao), KI3 (TaiXi), LR3 (TaiChong). All the acupoint were applied bilaterally.
  Laser divice directly contacts the points. All those points near the superficial roots of facial nerve. At each point, we treated for 1min, 1500 Hz, 50% laser intensity. And patients in PBMT group wore safety glasses to prevent eye damage during the laser sessions. All treatments were performed in the outpatient clinic by the same physician.
  Interventions: Device: Multiwave Locked System
- Control Group (Sham Comparator): Patients in the control group received no intervention but were free to pursue therapies if desired.
  Interventions: Device: Multiwave Locked System

INTERVENTIONS:
Device: Multiwave Locked System — Multiwave Locked System laser is a class IV NIR laser with two synchronized sources (905 nm with 75 W peak power, pulsed mode; 808 nm with power 1 W, continuous mode). Both laser beams were synchronized, the locked waves work with the range 1-2000 Hz.

SUMMARY:
OBJECTIVE: To determine whether photobiomodulation therapy by class IV Multiwave Locked System laser treatment could relieve symptoms in patients with Bell's palsy with a duration of greater than 8 weeks.

METHODS AND METHODS: This randomized controlled trial from May 2021 to April 2023. Patients were eligible who had Bell's palsy with a duration of greater than 8 weeks on out-patient department of otorhinolaryngology in Beijing Tongren Hospital. The photobiomodulation group received class IV Multiwave Locked System laser treatment for 3 times per weeks, a total of 6 months. The control group received the same Multiwave Locked System treatment procedure except the laser parameter. The primary outcome measures comprised House-Brackmann facial nerve grading system, Sunnybrook facial grading system, Facial Clinimetric Evaluation Scale. Secondary outcome measures comprised Electroneurography, Electromyography, and the Blink Reflex.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible for House-Brackmann grading system (HB) greater than or equal to grade 3.
* Patients were adults over 18 years of age and under 60 years of age;
* Patients were not received medicine before 2 weeks of trial, such as prednisolone.

Exclusion Criteria:

* Patients were excluded HB grade 6, or greater than 90% denervation on electroneuronography, or no voluntary electromyography activity, or no latency of early (R1) and late (R2, R2') components in Blink Reflex patients.
* Patients were excluded serious mental illness or social problems, and neurological disorders. And systemic disease, such as severe diabetes, malignant tumors, and other serious consumptive diseases, planning for pregnancy, in pregnancy or lactation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
House-Brackmann grading system | Change from Baseline number of pathological HB grading at 6-months in post-therapy.
  The House-Brackmann facial nerve grading system (HB grading) is based on a 6-grade score that offers a gross evaluation of facial motor function and includes the evaluation of sequelae. The prognoses of patients with House- Brackmann grade I or grade II were considered good, and the prognoses of those with grade 3 or higher were considered poor.
electroneuronography | Change from Baseline amplitude and potential of CAMP and the numbers of pathological ENoG at at 6-months in post-therapy.]
  The goal of the Electroneurography (ENoG) testing is to measure the amount of neural degradation that has occurred distal to the site of facial nerve injury by measuring the muscle response to an electrical stimulus. The testing of ENoG involves recording the compound muscle action potential (CAMP) of the mimetic muscles, including Orbicularis oculi, Frontalis muscle, Orbicularis oris and Zygomaticus muscle. ENoG is performed first on the healthy side of the face and then on the affected side. Nerve damage or nerve fiber degeneration leads to a decrease or loss of the CAMP. The amplitude of the CAMP on the affected side is compared to the CAMP of the healthy side and expressed as percent (amplitude of the paralyzed side divided by the amplitude of the normal side). A side difference of 30% or bigger is considered pathologic.

SECONDARY OUTCOMES:
Sunnybrook Facial Grading Scale | Change from Baseline number of pathological SB grading at 6-months in post-therapy.
  The Sunnybrook facial grading system (SB grading) is 13-items, self-reported questionnaire that used to evaluate the facial movement of patients. Among the overall 13 items of question, 3 items are resting symmetry, 5 items are symmetry of voluntary movement, and 5 items are synkinesis. Lower scores of Sunnybrook equate to greater severity of facial paralysis symptoms.
electromyography | Change from Baseline amplitude and duration of MUAPs at at 6-months in post-therapy.
  EMG is an electrophysiologic measures that indirectly quantify facial nerve function by recording motor unit action potentials (MUAPs) in the muscle of Musculus depressor angulli oris, Frontalis muscle and Orbicularis oris. MUAPs are the spikes in electrical activity generated when a motor unit fires. A motor unit consists of a motor neuron and the corresponding muscle fibers innervated by the neuron.
Blink Reflex | Change from Baseline number of pathological Blink Reflex at 6-months in post-therapy
  The blink reflex test is to measures the facial nerve since the blink reflex delivers information on facial nerve function with normal trigeminal function. Blink reflex testing involves electrical stimulation of the supraorbital nerve on the affected side combined with a 2-channel simultaneous sEMG recording from both orbicularis oculi muscles. The exit of the supraorbital nerve in the supraorbital foramen is palpated on the rim of the orbit. Stimulation with 10-20 mA and 0.2 ms duration is used to produce a constant reflex. In blink reflex testing, two responses, R1 and R2, are analyzed. R1 is the fast ipsilateral response of the orbicularis oculi muscle with a latency of about 10-12 ms. The second bilateral response R2 has a latency of about 30-41 ms.
  The R2 latency differences between both sides higher than 5-8 ms is considered pathologic.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing TongRen Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, Analytic Code

REFERENCES:
- [Derived] Wu D, Lan X, Litscher G, Zhao YL, Wu YQ, Dai RJ, Cao K, Wang Y, Chen LQ. Laser acupuncture and photobiomodulation therapy in Bell's palsy with a duration of greater than 8 weeks: a randomized controlled trial. Lasers Med Sci. 2024 Jan 13;39(1):29. doi: 10.1007/s10103-023-03970-4. PMID 38216803